CLINICAL TRIAL: NCT02376335
Title: B-Cell Depleting Therapy (Rituximab) as a Treatment for Fatigue in Primary Biliary Cirrhosis
Acronym: RITPBC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Department of Health, United Kingdom (Other Government); Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5997; 2012-000145-12 (EudraCT Number)
Record Dates: First submitted 2015-02-24; First posted 2015-03-03 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Fatigue; Primary Biliary Cirrhosis
Keywords: Fatigue; Primary Biliary Cirrhosis; Rituximab; PBC-40
MeSH Terms: conditions — Fatigue; Liver Cirrhosis, Biliary | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab infusion (Active Comparator): Participants will be randomised to Rituximab therapy (1000 mg IV on days 1 and 15) or placebo (0.9% Sodium Chloride 250mls) control.
  Interventions: Biological: Rituximab
- Placebo infusion (Placebo Comparator): Participants will be randomised to Rituximab therapy (1000 mg IV on days 1 and 15) or placebo (0.9% Sodium Chloride 250mls) control.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Rituximab — The Rituximab dosing regimen identified is that used in the proof of concept study, which is also the established treatment regimen for Rituximab use in rheumatoid arthritis. All interventions will be administered with a clinician present throughout the infusion in participants who have been encouraged to have adequate oral hydration in the 24 hours prior to attendance. Resuscitation equipment will be immediately available during the infusion period. Blood pressure, heart rate and temperature will be monitored during the infusion. Participants will continue to be observed in the Clinical Research Facility for at least 1 hour after the infusion.
  Other Names: MabThera
  Arms: Rituximab infusion
Other: Placebo — Participants will be randomised to Rituximab therapy (1000 mg IV on day 1 and 15) or placebo (0.9% Sodium Chloride 250 mls) control
  Other Names: 0.9% Sodium Chloride 250 mls
  Arms: Placebo infusion

SUMMARY:
Primary Biliary Cirrhosis (PBC) is a liver disease that predominantly affects females, can present for the first time at any age and which develops over many years. It is caused by the immune system attacking the body's own tissues. People with PBC frequently experience profound fatigue or tiredness which they liken to their "batteries running down" and although people still want to undertake normal activities they often lack the energy to be able to do them. This reduces quality of life, makes it difficult for people to work and can end up with them becoming isolated in the community. At present the investigators have no treatment for fatigue in PBC. Finding a treatment for fatigue in PBC is one of the highest research priorities identified by patient groups.

The aim of this study is to undertake a clinical trial to examine the effects of a treatment ("Rituximab") on severe fatigue in PBC to help us understand whether this will be a potentially useful treatment. The information that this will give us about how energy generation changes in patients with PBC with and without the treatment will also help us to develop new treatments for fatigue in other diseases. The study has the potential to improve the quality of life of many patients with PBC, for whom there is currently no hope of improvement.

The investigators will perform a randomised controlled study of Rituximab therapy in PBC compared to placebo (1:1 ratio).

The study will be performed in a specialised clinical research environment at Clinical Research Facility Royal Victoria Infirmary. The investigators have, for many years, worked closely with PBC patient groups to focus on the problems that are important to our patients. This study is fully supported by Liver North, a liver disease charity and patient support group.

The study will take place over one year and will involve between 9 and 20 visits although a number of these will be telephone visits. Blood tests and quality of life questionnaires will be performed at the start of the study and after three, six, nine and twelve months. At baseline and 12 weeks follow up physical activity will be monitored using monitors, and an exercise test and MRI scan will be performed.

DETAILED DESCRIPTION:
Primary Biliary Cirrhosis (PBC) is a liver disease that predominantly affects females, can present for the first time at any age, and which develops over many years. It is caused by the immune system attacking the body's own tissues. People with PBC frequently experience profound fatigue or tiredness which they liken to their "batteries running down", and although people still want to undertake normal activities they simply lack the energy to be able to do them. This reduces quality of life, makes it difficult for people to work, and can end up with them becoming isolated in the community. At present we have no treatment for fatigue in PBC. Finding a treatment for fatigue in PBC is one of the highest research priorities identified by patient groups.

We have shown that PBC patients with fatigue have an abnormality in the way they generate energy within their muscles. This appears to be associated with the presence of an antibody in the blood which is directed against an important protein which normal cells in the body use to generate energy. In recent years new drug treatments have been developed which allow us to safely suppress the part of the immune system which produces antibodies of the type that seem to cause energy production problems in PBC. As yet, however, the extent to which these medicines can improve fatigue through removal of antibodies in PBC has not been tested.

The aim of this study is to undertake a clinical trial to examine the effects of this treatment ("Rituximab") on severe fatigue in PBC to help us understand whether this will be a potentially useful treatment. This will give us information about how energy generation changes in patients with PBC and will also help us to develop new treatments for fatigue in other diseases. The study has the potential to improve the quality of life of many patients with PBC, for whom there is currently no licensed treatment.

We will perform a randomised controlled trial of Rituximab therapy in PBC compared to placebo with the primary end point of fatigue severity. The study will be performed in a specialised PBC clinical centre.

Our hypothesis is that the B-cell-directed immunotherapeutic agent Rituximab will improve fatigue in PBC (an important and disabling symptom) through its effect on B-cells producing antibodies which inhibit the function of pyruvate dehydrogenase (PDH) an important energy generating enzyme.

Fatigue is a common and debilitating symptom which frequently impacts significantly on quality of life and ability to function in patients with PBC. There are currently no effective treatments for fatigue in PBC and new approaches are urgently required to address this unmet need. Rituximab, a B-cell depleting agent, holds specific promise (with evidence from a small-scale proof-of-concept pilot trial) as a therapy for fatigue in PBC, given the strong evidence linking the antibody response to PDH in the pathogenesis of fatigue in this disease. We also believe, given the robust diagnostic criteria and the availability of validated clinical tools, that PBC is an important and useful human model in which to study the pathogenesis and treatment of fatigue.

There are currently no treatments for fatigue in PBC and we are not aware of any other treatments under evaluation.

A pilot study performed in Canada exploring the use of Rituximab in PBC (in 13 patients) has provided proof-of-concept, showing that the agent is safe and well-tolerated in patients, and is associated with a clinically significant reduction in fatigue. Fatigue severity was assessed using the Fatigue Severity Scale (FSS) (potential range 9-63 points) with a fall being seen from pre-treatment (median FSS=36, range 11-59) to post-treatment (median=29, range 12-55). Taking into account the floor value for the FSS, this represents a median fall in fatigue severity over 6 months of 26%. This compares with our own case-control study of fatigue in PBC which suggests that fatigue severity in age and sex matched normal controls is 30% lower than in PBC patients1 suggesting the potential for Rituximab therapy to return PBC patients to close to normal with regards to their perceived fatigue. However, this pilot study did not attempt to explore the mechanism of the effect, and since it did not use severe fatigue as an inclusion criteria, the extent of possible improvement for such patients is unclear; moreover, the study was not optimised for the study of fatigue (fatigue was a secondary outcome and only some of the patients who participated had fatigue potentially under-estimating the clinical effect). Patients showed a sustained reduction in anti-PDH antibody levels of all isotypes, supporting the concept that Rituximab has a beneficial effect on fatigue through depletion of PDH-reactive antibody.

The importance of severe fatigue in PBC and the current lack of treatments, the strong theoretical basis for the approach, and the supportive pilot trial proof-of-concept data all, we believe, justify a formal clinical trial of Rituximab targeting fatigue in PBC. Data from animal models of PBC implicating activated B-cells in promoting autoreactivity, from human in vitro studies showing increased TLR-mediated B-cell activation in PBC, from human genetic studies showing disease associations with loci implicated in regulation of the B-cell pool size and the pilot trial data showing improvement in liver biochemistry in PBC patients treated with Rituximab all point to the potential for an additional, more generic benefit for this treatment in terms of underlying liver inflammation further justifying a substantive clinical trial in PBC.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* patient has capacity and provided written informed consent for participation in the study prior to any study specific procedures
* moderate or severe fatigue as assessed using previously designated cut-offs of the PBC-40 fatigue domain (i.e. fatigue domain score >33)
* presence of AMA (anti-PDH antibody) at a titre of >1:40
* adequate haematological function Hb >9g/L, Absolute neutrophil count >1.5x109/L, platelet count > 50x109/L
* bilirubin ≤ 50 μmol
* INR ≤ 1.5
* Child-Pugh score < 7
* ECOG performance status < 2
* adequate renal function; Cockroft and Gault estimation > 40ml/min
* women of childbearing potential should have a negative pregnancy test prior to study entry AND be using an adequate contraception method, which must be continued for 12 months after completion of treatment. Acceptable forms of effective contraception include:

  * established use of oral, injected or implanted hormonal methods of contraception
  * placement of an intrauterine device (IUD) or intrauterine system (IUS)
  * barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository
  * male sterilisation (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate)
  * true abstinence: when this is in line with the preferred and usual lifestyle of the subject

Exclusion Criteria:

* advanced or decompensated disease (variceal bleed, hepatic encephalopathy or ascites)
* history or presence of other concomitant liver diseases (including hepatitis due to hepatitis B (surface antigen positive or core antibody positive) or C or evidence of chronic viraemia on baseline screening), primary sclerosing cholangitis or biopsy proven non-alcoholic steatohepatitis)
* average alcohol ingestion >21 units/week (male) or >14 units / week (female)
* chronic sepsis or intercurrent condition likely to predispose to chronic sepsis during the study
* previous treatment with B-cell depleting therapy
* previous history of aberrant response or intolerance to immunological agents
* presence of significant untreated intercurrent medical condition itself associated with fatigue
* presence of significant risk of depressive illness (HADS score indicating caseness)
* current statin therapy or statin use within 3 months of enrolment
* ongoing participation in other clinical trials or exposure to any investigational agent 4 weeks prior to baseline or within < 5 half lives of the investigational drug
* major surgery within 4 weeks of study entry
* vaccination within 4 weeks of study entry; patients requiring seasonal flu or travel vaccines will be required to wait a minimum of 4 weeks post vaccination to enrol in the study
* pregnant or lactating women
* psychiatric or other disorder likely to impact on informed consent
* patient is unable and/or unwilling to comply with treatment and study instructions
* any other medical condition that, in the opinion of the investigator would interfere with safe completion of the study
* hypersensitivity to the active substance (Rituximab) or to any of the excipients (sodium citrate, polysorbate 80, sodium chloride, sodium hydroxide, hydrochloric acid, water (for infusion)) or to murine proteins
* active, severe infections (e.g. tuberculosis, sepsis or opportunistic infections)
* known HIV infection
* clinical history of latent TB infection unless the patient has completed adequate antibiotic prophylaxis
* AST/ALT 4 x upper limit of normal
* severe immune-compromised state
* severe heart failure (NYHA Class IV) or severe uncontrolled cardiac disease
* malignancy (other than basal cell carcinoma) within the last 10 years
* demyelinating disease
* previous participation in this study
* any contraindication to Rituximab therapy not covered by other exclusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-10; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Fatigue severity in PBC patients, assessed using the fatigue domain of the PBC-40, a fully validated, psychometrically robust, disease specific quality of life measure | Between baseline and 12 week assessment

SECONDARY OUTCOMES:
Improvement in physical activity assessed using seven day physical activity monitoring | 12 weeks
Assessment of improvement in daytime somnolence, vasomotor autonomic symptoms, functional status, reduction in depressive and anxiety-related symptoms | 12 weeks
  All assessments will be using questionnaires that currently are used in the routine clinical setting.
Reduction in serum anti-pyruvate dehydrogenase complex antibody levels and in numbers of peripheral blood B-cells | 12 months
  This is to confirm whether any clinical effect is directly related to antibody modulation.
Improvement in peripheral muscle bio-energetic function on exercise | 12 weeks
  This is to confirm whether any clinical effect is directly related to effects on muscle bioenergetic function.

CONTACTS AND LOCATIONS:
Overall Officials: David EJ Jones, BA, BM, MRCP, PhD, FRCP, Principal Investigator — Faculty of Medical Sciences, Newcastle University
Locations (1):
- Newcastle Clinical Trials Unit, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- [Derived] Khanna A, Jopson L, Howel D, Bryant A, Blamire A, Newton JL, Jones DE. Rituximab Is Ineffective for Treatment of Fatigue in Primary Biliary Cholangitis: A Phase 2 Randomized Controlled Trial. Hepatology. 2019 Nov;70(5):1646-1657. doi: 10.1002/hep.30099. Epub 2018 Sep 22. PMID 29790196